CLINICAL TRIAL: NCT04808245
Title: A MultIceNTER Phase I Peptide VaCcine Trial to Exploit NeoePitope-Specific T Cells for the Treatment of H3-Mutated Gliomas - (INTERCEPT-H3)
Brief Title: A MultIceNTER Phase I Peptide VaCcine Trial for the Treatment of H3-Mutated Gliomas
Acronym: INTERCEPT-H3
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Charite University, Berlin, Germany (Other); Roche Pharma AG (Industry); German Cancer Aid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2018-576
Record Dates: First submitted 2021-03-05; First posted 2021-03-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Newly Diagnosed H3-mutated Glioma
Keywords: Diffuse midline glioma; Histone H3; H3K27M; DIPG; Glioma; Glioblastoma; Immunotherapy
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — atezolizumab; Injections; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard patient cohort (Experimental): All fifteen patients will receive in total 11 doses of H3K27M peptide vaccine starting with standard radiotherapy (RT) and 14 doses of the human anti-PD-L1 antibody Atezolizumab/ Tecentriq® (every three weeks, q3w) starting four weeks after completion of RT. The first 3 vaccines will be given bi-weekly (q2w) in combination with RT. One dose of vaccination will be given at the beginning of recovery (RE) period following RT. Vaccines 5-11 (q6w) will be initiated with Atezolizumab after completion of RE. The H3K27M peptide vaccine is administered in combination with topical Imiquimod that serves as an adjuvant.
  For safety reasons, the first three patients will be enrolled sequentially: Each patient will receive the first vaccination at the earliest 28 days after the previous patient has received the first vaccination.
  Interventions: Drug: Tecentriq 1200 MG in 20 ML Injection; Biological: H3K27M peptide vaccine; Other: Imiquimod (5%)

INTERVENTIONS:
Drug: Tecentriq 1200 MG in 20 ML Injection — One vial of Tecentriq® (1200 mg) will be administered as an intravenous (i.v.) infusion over 60 minutes every 3 weeks starting 4 weeks after radiotherapy. If the first infusion is tolerated, all subsequent infusions will be delivered over 30 minutes.
  Other Names: Atezolizumab
Biological: H3K27M peptide vaccine — The H3K27M peptide vaccine is injected subcutaneously (s.c.). For a single vaccination 300 μg of the peptide will be emulsified in a total volume of 1 ml.
Other: Imiquimod (5%) — One sachet of Aldara® cream (250 mg) will be applied to an area of 5 x 5 cm around the injection site of the H3K27M peptide vaccine 15 min after vaccination and left on the skin for approximately 8 hours according to the instructions in the SmPC. 24 hours after the vaccination a second sachet of Aldara® will be applied by the patient as instructed above and left on the skin for approximately 8 hours.
  Other Names: Aldara

SUMMARY:
The study "A MultIceNTER Phase I Peptide VaCcine Trial to Exploit NeoePitope-Specific T Cells for the Treatment of H3K27M-Mutated Gliomas - (INTERCEPT H3)" is a non-controlled, open-label, single arm, multicenter phase I trial involving patients with gliomas carrying an H3.1K27M or H3.3K27M mutation.

DETAILED DESCRIPTION:
The patient population will be molecularly defined and include adult patients with newly diagnosed K27M-mutant histone-3.1 (H3.1K27M) or histone-3.3 (H3.3K27M) diffuse midline gliomas (DMG).

Within this trial, a long peptide vaccine containing a K27M-mutated histone-3 sequence, will be administered subcutaneously in addition to standard radiotherapy and thereafter in combination with the human anti-PD-L1 antibody Atezolizumab.

Fifteen patients (pts. 1-15) will receive 11 doses of H3K27M peptide vaccine in total starting with standard radiotherapy (RT) and 14 doses of the human anti-PD-L1 antibody Atezolizumab (every three weeks, q3w) starting four weeks after completion of RT. The first 3 vaccines will be given bi-weekly (q2w) in combination with RT. One dose of vaccination will be given at the beginning of recovery (RE) period following RT. Vaccines 5-11 (q6w) will be initiated with Atezolizumab after completion of RE. In a safety lead-in, the first three patients (pts. 1-3) will be enrolled sequentially.

Following the last IMP administration, a safety / immunogenicity follow-up is planned for 24 weeks until end of study (EOS). To be able to assess safety, tolerability and immunogenicity of the peptide vaccine in combination with Atezolizumab 15 evaluable patients will be enrolled.

Diffuse gliomas of the thalamus, brain stem, spinal cord or other midline structures represent 3-4% of high-grade glioma and harbor H3.1K27M or H3.3K27M mutations as a characteristic founder mutation in > 70% of cases. H3K27M-mutant gliomas typically occur in children and adolescents but also in adult patients. After biopsy or resection, the standard of care consists of involved-field radiotherapy. Adding alkylating chemotherapy to radiotherapy does not offer additional benefit in retrospective case series and prospective clinical trials in children with pontine gliomas, probably as hypermethylation of the MGMT promoter in DMG is typically lacking. After radiotherapy gliomas frequently recur with a median 12-month progression-free survival of 20 %. Importantly, at recurrence particularly in the adult patient population, there is frequent distant progression and leptomeningeal dissemination, arguing for the necessity of systemic therapy upfront.

From an immunological point of view H3K27M represents an attractive tumor antigen specifically expressed in tumor but not normal cells. Patients with H3K27M-mutant gliomas may harbor mutation-specific T cells, indicating that H3K27M is specifically presented to and recognized by the immune system in a mutation-specific manner. Vaccination of humanized mice with a long H3K27M vaccine results in an anti-tumor immune response effective in controlling H3K27M-expressing tumors in a preventive and a therapeutic manner without causing toxicity. In addition, eight adult patients with H3.3K27M-mutated gliomas were treated with an H3K27M 27 amino acid long peptide vaccine on a compassionate-use basis. None of the patients treated either with the peptide vaccine alone or in combination with an anti-human PD(L)-1 antibody showed any clinical or laboratory sign of treatment-related toxicity except for grade 1 injection site reactions. Importantly, all patients developed H3K27M-specific T cell responses with one patient of the combination treatment group showing long-term response with no sign of tumor progression for >24 months after vaccination and one patient experiencing complete response after pseudoprogression (unpublished observations). Based on these observations we hypothesize that checkpoint inhibition targeting PD-L1 is required for optimal amplification of a vaccine-induced H3K27M-specific T cell response.

The aim of this phase I trial is to evaluate the safety and immune response to the H3K27M peptide vaccine in combination with Atezolizumab in patients with H3K27M-mutant diffuse midline gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients present with histologically confirmed diagnosis of an H3.1K27M or H3.3K27M-mutated diffuse midline glioma WHO grade IV (with or without measurable residual tumor after tumor resection or biopsy after primary diagnosis)
* Tumoral H3.1K27M or H3.3K27M mutation proven by immunohistochemistry or H3 DNA sequencing
* No previous treatment except for surgery
* Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Availability of tumor tissue for translational analyses (FFPE bulk tissue or biopsy)
* Patients are scheduled to receive radiotherapy
* Patients should be immunocompetent (i.e. no concomitant treatment with dexamethasone (or equivalent), or receive stable/decreasing steroid levels not exceeding 2 mg/day dexamethasone (or equivalent) during the last 3 days prior to clinical screening; no severe lymphopenia)
* minimum 18 years old, smoking or non-smoking, of any ethnic origin and sex
* Karnofsky Performance Status minimum 60. For patients with spinal gliomas, paralysis-caused mobility impairments will not be considered
* Ability of patient to understand character and individual consequences of the clinical trial
* Evidence of informed consent document personally signed and dated by the patient (or a witness in case the patient is unable to write) covering all trial-related procedures and indicating that the patient has been informed of all pertinent aspects of the study and that the patient consents to participate in the trial.
* Non-nursing and non-pregnant women: Women of child-bearing potential (WOCBP) must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) prior to the start of the investigational medicinal product (IMP). A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In case of possible postmenopausal status or doubtful childbearing potential, assessment of serum FSH (follicle-stimulating hormone) level will be performed once at baseline visit to confirm postmenopausal status. In this case, urine pregnancy tests during the trial as well as contraception are not necessary. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* WOCBP must be using a highly effective method of birth control (failure rate of less than 1% per year) to avoid pregnancy throughout the study and at least 5 months after the last dose of the IMP. Such methods include:

  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral intravaginal transdermal
  * progestogen-only hormonal contraception associated with inhibition of ovulation: oral injectable implantable
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system (IUS)
  * bilateral tubal occlusion
  * vasectomised partner
  * sexual abstinence
* Fertile men must be willing and able to use an effective method of birth control (condom) throughout the study for up to at least 5 months after the last dose of the IMP, if their sexual partners are WOCBP, using an effective method as well (acceptable methods see above). A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Current use of immunosuppressive medication including treatment with systemic immunomodulatory agents at least 4 weeks or five half-lives of the drug, prior to starting study treatment, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Previous or concurrent standard or experimental treatment for the tumor other than resection. This includes local therapies such as interstitial radiotherapy or local chemotherapy (i.e. BCNU wafers), loco-regional hyperthermia, electric fields, and antiangiogenic therapy (such as Bevacizumab).
* Abnormal (≥ Grade 2 CTCAE v5.0) laboratory values for thyroid gland: free T4 and TSH
* Abnormal (≥ Grade 2 CTCAE v5.0) laboratory values for hematology, liver and renal function (serum creatinine). In detail, the following values apply as exclusion criteria:

  1. Hemoglobin < 9 g/dL (5.59 mmol/L)
  2. White blood cell count (WBC) decrease (<3.0 x 109/L) or increase (> 10.0 x 109/L)
  3. Absolute neutrophil count (ANC) decrease (< 1.5 x 109/L)
  4. Platelet count decrease (< 100 x 109/L)
  5. Bilirubin > 1.5 x ULN (upper limit of normal according to the performing lab´s reference range)
  6. ALT > 2.5 x ULN
  7. AST > 2.5 x ULN
  8. GGT > 2.5 x ULN
  9. Serum creatinine increase (> 1.5 x ULN)
* Patients with history or presence of HIV and/or HBV/HCV positivity (testing performed according to local standards)
* Patients with history or known presence of tuberculosis (positive QuantiFERON®-TB Gold test or tuberculin skin test). Patients with an indeterminate result of the QuantiFERON®-TB Gold test are not eligible unless additional testing demonstrates a negative result (tuberculin skin test or repeated QuantiFERON®-TB Gold test). If a tuberculin skin test is performed, an induration of > 6 mm is "positive" for a patient with history of BCG vaccine, while an induration of > 10 mm is "positive" for a patient without history of BCG vaccine. If necessary, a QuantiFERON®-TB Gold test might be complemented by additional specific diagnostic tests as per standard procedures.
* Patients with severe infection(s) or signs/symptoms of infection within 2 weeks prior to start of treatment including radiotherapy and IMP
* Active infection requiring systemic therapy
* Patients who have received a live, attenuated vaccine within 4 weeks prior to start of treatment including radiotherapy and IMP
* Patients with a prior solid organ transplantation or hematopoietic stem cell transplantation
* Active autoimmune disease including history of severe autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible
* Clinically significant (i.e. active) cardiovascular disease: Cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 5 years unless the patient has been diseasefree for 5 years.
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3)
* Participation in other clinical trials or their observation period during the last 30 days before start of treatment including radiotherapy and IMP

No patient will be allowed to enroll in this trial more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety of repeated fixed dose vaccinations with the H3K27M peptide vaccine administered with radiotherapy and Atezolizumab in patients with H3K27M-mutant gliomas. Primary safety endpoint is the Regime Limiting Toxicity (RLT). | Through study completion, an average of one year
  Safety of H3K27M peptide vaccine administered with radiotherapy and Atezolizumab. Primary safety endpoint is the Regime Limiting Toxicity (RLT).
Assessment of immunogenicity of repeated fixed dose vaccinations with the H3K27M peptide vaccine administered with radiotherapy and Atezolizumab in patients with H3K27M-mutant gliomas. | From Day 1 until the date of study termination (until day 540); approximately 16 times
  Immunogenicity (Immune response Yes/No) will be assessed for all evaluable patients. The primary immunogenicity endpoint is the presence of an H3K27M-specific T-cell response. H3K27M-specific T cell responses are measured on Peripheral Blood Mononuclear Cells (PBMC) using IFN-gamma ELISpot.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From day of first diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to the date of study termination (approximately until day 540)
  PFS, defined as time from the day of first diagnosis to the day of local tumor progression or the day of death of any cause (whichever occurs first), censored by the end of the observation. PFS analysis will be based on the central disease assessment (refer to section 7.5.1). Patients lacking an evaluation of tumor response (based on radiological or clinical assessment) will have their PFS time censored on the date of first diagnosis with duration of 1 day.
Overall response rate (ORR) | Baseline visit to end of study (approximately until day 540)
  ORR, defined as the proportion of patients showing complete response (CR), partial response (PR) or stable disease (SD) at EOS compared to the baseline value (MRI at visit 1 for ORR under trial drug). ORR analysis will be based on the central disease assessment according to the iRANO criteria.
Analyze the association between immunogenicity and the clinical outcome parameters ORR | Through study completion, an average of one year
Analyze the association between immunogenicity and the clinical outcome parameters PFS | Through study completion, an average of one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Platten, Prof., Principal Investigator — German Cancer Research Center Germany
Locations (8):
- Germany (8):
  - Department of Neurology and Polyclinic, Universitiy Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Medical Center Mannheim, Department of Neurology, Mannheim, Baden-Wurttemberg
  - University Clinic Tuebingen, Neurological Clinic, Department of Neurology, Tübingen, Baden-Wurttemberg
  - Dr. Senckenberg Institute for Neurooncology, University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Clinical Neuro-Oncology Section, University Hospital Bonn (UKB), Bonn, North Rhine-Westphalia
  - Neurooncology Department, University Hospital Essen, Essen, North Rhine-Westphalia
  - Clinic and Polyclinic for Neurosurgery, University Hospital Carl Gustav Carus Dresden, Dresden, Saxony
  - Department of Neurosurgery with Pediatric Neurosurgery, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ochs K, Ott M, Bunse T, Sahm F, Bunse L, Deumelandt K, Sonner JK, Keil M, von Deimling A, Wick W, Platten M. K27M-mutant histone-3 as a novel target for glioma immunotherapy. Oncoimmunology. 2017 May 12;6(7):e1328340. doi: 10.1080/2162402X.2017.1328340. eCollection 2017. PMID 28811969
- [Derived] Grassl N, Sahm K, Susse H, Poschke I, Bunse L, Bunse T, Boschert T, Mildenberger I, Rupp AK, Ewinger MP, Lanz LM, Denk M, Tabatabai G, Ronellenfitsch MW, Herrlinger U, Glas M, Krex D, Vajkoczy P, Wick A, Harting I, Sahm F, von Deimling A, Bendszus M, Wick W, Platten M. INTERCEPT H3: a multicenter phase I peptide vaccine trial for the treatment of H3-mutated diffuse midline gliomas. Neurol Res Pract. 2023 Oct 19;5(1):55. doi: 10.1186/s42466-023-00282-4. PMID 37853454